CLINICAL TRIAL: NCT01109979
Title: Effect of Combined Estradiol and Drospirenone Treatment Versus Combined Estradiol and Medroxyprogesterone Acetate Treatment on Endothelial Function: A Crossover Study
Brief Title: Effect of Estradiol+Drospirenone Versus Estradiol+MPA on Endothelial Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Ellen W. Seely, M.D., Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 2006p002137
Record Dates: First submitted 2010-04-22; First posted 2010-04-23 (Estimated); Results first posted 2013-05-03 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-06

CONDITIONS: Cardiovascular Diseases
Keywords: Cardiovascular, vascular
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Lunelle; drospirenone and ethinyl estradiol combination; estradiol-drospirenone combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Estradiol+MPA (Active Comparator)
  Interventions: Drug: Estradiol+MPA
- Estradiol+DRSP (Active Comparator)
  Interventions: Drug: Estradiol+Drospirenone

INTERVENTIONS:
Drug: Estradiol+MPA — 1 single pill dose daily containing estradiol 1 mg + medroxyprogesterone acetate 2.5 mg
  Other Names: Estradiol+medroxyprogesterone acetate
  Arms: Estradiol+MPA
Drug: Estradiol+Drospirenone — 1 single pill dose daily containing estradiol 1mg + drospirenone 0.5 mg
  Other Names: Angeliq
  Arms: Estradiol+DRSP

SUMMARY:
This study compares the effects of two common hormone medications on the heart and blood vessels of healthy post-menopausal women over the age of 45.

The study will take place over the course of about 5 months. Each subject will take two different medications over two six-week periods. They will be randomized at the beginning of the study to either estradiol+medroxyprogesterone acetate or estradiol+drospirenone for the first period, and will receive the other medication the second six-weeks of the study. At the very beginning of the study and at the end of each six-week treatment period, subjects will come to the hospital various tests including non-invasive blood vessel imaging tests, blood draws to test the levels of certain hormones in the body, an oral glucose tolerance test, a test to monitor renal blood flow, and 24-hour blood pressure monitoring. Between treatment periods, there will be a four-week medication-free washout period.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female postmenopausal volunteers, as defined by absence of menses for at least 12 months and follicle stimulating hormone (FSH) 30 IU/L;
2. Age 45 to 75 years;
3. Systolic blood pressure <140 and >90 mmHg and diastolic blood pressure <90 and >60 mmHg at the screening visit;
4. No personal history of diabetes;
5. Body mass index < 30 kg/m2;
6. No clinically significant abnormalities on screening tests (complete blood count, serum electrolytes, liver enzymes, thyroid stimulating hormone, urinalysis, and electrocardiogram).

Exclusion Criteria:

1. Current smoking, defined as smoking within the 12 months before the screening visit;
2. Alcohol intake >1 beverage per night or history of alcohol abuse;
3. Current or past recreational drug use;
4. Personal history of hypertension, cardiovascular disease (coronary artery disease, congestive heart failure, valvular heart disease, stroke, transient ischemic attack, or intermittent claudication), hyperlipidemia, diabetes (defined as a fasting glucose ≥126 mg/dL), kidney disease, liver disease, venous or arterial thromboembolic disease, adrenal insufficiency, depression, or illness requiring overnight hospitalization in the past 6 months;
5. Risk factors for arterial or venous thromboembolism;
6. Personal history of breast cancer or any other type of cancer;
7. Personal history of endometrial hyperplasia, endometrial cancer, or unexplained vaginal bleeding;
8. History of cervical cancer or abnormal pap smear
9. Prescription or herbal medication use, excluding thyroid hormone supplementation;
10. Ischemic changes on resting electrocardiogram;
11. Serum creatinine ≥ 1.3 mg/dL.
12. Serum potassium level > 5.0 mmol/L;
13. Known hypersensitivity to any of the study drugs;
14. Other active medical problems detected by examination or laboratory testing, except for treated hypothyroidism.
15. Pregnancy

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-12; Primary Completion 2012-01 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Seely, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Postmenopausal women ages 45 and 75 were recruited 2009- 2011 via flyers, newspaper advertisements, Craigslist, RSVP for Health, and websites.
Pre-assignment Details: Subjects were excluded after screening procedures due to history of hypertension, cardiovascular disease, hyperlipidemia, diabetes, liver disease, cancer, elevated creatinine/potassium levels, abnormal thyroid function, and evidence that menopause was not completed.
Groups:
- E+MPA, Then E+DRSP: Estradiol (E) 1 mg orally per day + medroxyprogesterone acetate (MPA) 2.5 mg orally per day for 6 weeks, then 4 week washout before Estradiol (E) 1 mg orally per day + Drospirenone (DRSP) 0.5 mg orally per day for 6 weeks
- E+DRSP, Then E+MPA: Estradiol (E) 1 mg orally per day + Drospirenone (DRSP) 0.5 mg orally per day for 6 weeks, then 4 week washout before Estradiol (E) 1 mg orally per day + medroxyprogesterone acetate (MPA) 2.5 mg orally per day for 6 weeks
Period: Overall Study
Arm/Group | E+MPA, Then E+DRSP | E+DRSP, Then E+MPA
Started | 12 | 12
Completed | 10 | 11
Not Completed | 2 | 1
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | E+MPA, Then E+DRSP | E+DRSP, Then E+MPA | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 10 | 18
  >=65 years | 4 | 2 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 12 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 11 | 10 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Brachial Artery Reactivity % Flow Mediated Dilation (BAR %FMD)
Description: This crossover study examined the effects of E+MPA versus E+DRSP on brachial artery reactivity (BAR) assessed after six weeks of treatment. BAR is a noninvasive measure of endothelium-dependent flow-mediated vasodilation (FMD) of the brachial artery. With this technique, inflation of an arm blood pressure cuff to suprasystolic blood pressure causes relative ischemia downstream to the cuff. Upon deflation, a brief state of increased blood flow occurs (reactive hyperemia), and the resulting increase in shear stress causes nitric oxide release and resulting vasodilation of the brachial artery (flow-mediated vasodilation). The flow-mediated changes in brachial artery diameter can be imaged by ultrasound and measured as an index of peripheral vasomotor function. BAR correlates with invasive assessments of coronary endothelial function as well as multiple cardiovascular risk factors.
Time Frame: %FMD after 6 weeks of treatment
Population: The number of participants for analysis includes only the participants that completed a baseline assessment and at least one of the treatment arms.
Measure: Mean (Standard Deviation); unit: % FMD after 6 weeks of treatment
Groups:
- E+MPA: Estradiol (E) 1 mg orally per day + medroxyprogesterone acetate (MPA) 2.5 mg orally per day for 6 weeks
- E+DRSP: Estradiol (E) 1 mg orally per day + Drospirenone (DRSP) 0.5 mg orally per day for 6 weeks
Arm/Group | E+MPA | E+DRSP
Number analyzed (Participants) | 21 | 21
% FMD after 6 weeks of treatment | 5.49 (3.32) | 3.39 (3.18)
Statistical Analysis 1: Comparison: E+MPA vs E+DRSP; Test type: Superiority or Other; p = 0.04, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | E+MPA | E+DRSP
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24

LIMITATIONS AND CAVEATS:
There may have been an order effect of E+DRSP on FMD. For this, however, we would expect %FMD to be lower in the 2nd treatment period, regardless of specific treatment. It is unclear whether this was true cross-over effect or due to the study size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No